CLINICAL TRIAL: NCT05723991
Title: Evaluation of an Open, Single Arm, Multicenter Phase II Clinical Study on the Neoadjuvant Treatment of HER2 Expressing Myometrial Invasive Bladder Cancer With Disitamab Vedotin for Injection and Gemcitabine
Brief Title: Study of Disitamab Vedotin Combined With Gemcitabine in Neoadjuvant Treatment of Urothelial Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunguang yang (101937) (Other)
Responsible Party: Sponsor-Investigator, Chunguang yang (101937), Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [222] LSZ (S137) No
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Radical Cystectomy; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — disitamab vedotin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vidiximab and Gemcitabine Neoadjuvant therapy (Experimental): Vidiximab (RC48) 2.0mg/kg, once every two weeks, intravenous drip (60-90 min); Gemcitabine is 1000mg/m2, once every 2 weeks
  Interventions: Drug: Disitamab Vedotin and Gemcitabine

INTERVENTIONS:
Drug: Disitamab Vedotin and Gemcitabine — Disitamab Vedotin (RC48) 2.0mg/kg, once every two weeks, intravenous drip (60-90 min); Gemcitabine is 1000mg/m2, once every two weeks. After completing 3 cycles of neoadjuvant combined therapy, imaging evaluation was performed. If the tumor is T0, radical surgery for bladder cancer was performed; Otherwise, perform radical surgery for bladder cancer after completing 1-3 cycles of treatment (total cystectomy+standard/extended lymph node dissection)

SUMMARY:
A multicenter, open, single arm, phase II clinical trial was designed for myometrial invasive bladder cancer to evaluate the efficacy and safety of RC48-ADC combined with gemcitabine in preoperative neoadjuvant treatment of MIBC, and provide high-level clinical evidence for gemcitabine combined with ADC in the treatment of MIBC

DETAILED DESCRIPTION:
Patients with myometrial invasive bladder cancer expressing HER2 and not suitable for cisplatin chemotherapy were treated with vedixizumab (RC48) 2.0mg/kg, once every two weeks, intravenous drip (60-90min); Gemcitabine is 1000mg/m2, once every two weeks. After completing 3 cycles of neoadjuvant combined therapy, imaging evaluation was performed. If the tumor is T0, radical surgery for bladder cancer was performed; Otherwise, perform radical surgery for bladder cancer (total cystectomy+standard/extended lymph node dissection) after completing 1-3 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study, signed the informed consent form, and were able to follow the study and follow-up procedures
2. Age 18-75
3. Suitable and planned for radical cystectomy (including lymph node dissection)
4. Clinical stage T2-T4aN0M0 (CT/MR/PET-CT evaluation)
5. Pathologically, it is urothelial carcinoma, and the patient has HER2 expression and refuses neoadjuvant chemotherapy or physical condition/renal function [glomerular filtration rate (GFR) 30-60mL/min], which is not suitable for neoadjuvant chemotherapy (pathology allows urothelial carcinoma to merge with other variant subtypes, with urothelial carcinoma as the main type)
6. ECOG score 0 or 1
7. There is residual tumor after TURBT (cystoscopy or imaging evidence)
8. The blood test of subjects should meet the following requirements

Exclusion Criteria:

1. Receive live attenuated vaccine within 4 weeks before enrollment or during the study period.
2. Have received systemic chemotherapy and targeted therapy of anti-PD-1, PD-L1 and HER2 in the past 6 months
3. Known allergy to gemcitabine/RC48 and its components
4. Active, known or suspected autoimmune diseases.
5. A history of primary immunodeficiency is known.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-09-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | three years
  Neoadjuvant therapy and postoperative pathology confirmed that the primary tumor was in complete remission (stage ypT0) and had no residual tumor cells, regardless of whether the regional lymph nodes were involved or not.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiquan hu, doctor, Study Director — Tongji Hospital
Locations (2):
- China (2):
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No